CLINICAL TRIAL: NCT01864668
Title: the Influence of Different Tidal Volume to Lung Strain of ARDS Patients
Brief Title: the Influence of Tidal Volume to Lung Strain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Xiaohua Qiu, physician, Zhongda Hospital
Other Study IDs: 20130519
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-05

CONDITIONS: Critically Ill; Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; lung strain; small tidal volume
MeSH Terms: conditions — Critical Illness; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Measure the lung strain in different tidal volume in ADRS patients to find the relationship between tidal volume and lung strain and find the most suitable tidal volume for each patient.

DETAILED DESCRIPTION:
Purpose:Find the relationship between tidal volume and lung strain in ARDS patients.Then find the most suitable tidal volume for each patient according to the dividing value.

Methods:Measure the lung strain in the tidal volume of 6mL/kg,8mL/kg,10mL/kg and 12mL/kg in each ARDS patient.

Hypothesis:With the increase of the tidal volume,the lung strain develops.In the patient with larger lung compliance,the strain of the group of conventional tidal volume is less than 0.27 and there is no obvious difference between the group of small tidal volume.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-85,gender is not limited
2. Needing Invasive ventilation
3. Fit the definition of ARDS in 2012 "Berlin Definition"
4. Sign the paper of informed consent

Exclusion Criteria:

1. pregnancy and at the end stage of tumour
2. the COPD patients
3. less than 24h of mechanical ventilation
4. more than 5 days of mechanical ventilation
5. FiO2>80%
6. presence of air leaks
7. organ dysfunction and hemodynamic instability
8. including in other research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients diagnosed with acute respiratory distress syndrome
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the strain in different tidal volume | 2 hours
  Use the GE ventilator to measure the EELV and calculate the lung strain(lung strain = VT/EELV)

SECONDARY OUTCOMES:
28 days mortality | 28 days
  Follow up to determine the mortality in 28 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xie J, Jin F, Pan C, Liu S, Liu L, Xu J, Yang Y, Qiu H. The effects of low tidal ventilation on lung strain correlate with respiratory system compliance. Crit Care. 2017 Feb 3;21(1):23. doi: 10.1186/s13054-017-1600-x. PMID 28159013